CLINICAL TRIAL: NCT00665717
Title: The Influence of Raltegravir on Pravastatin Pharmacokinetics in Healthy Volunteers (GRAPPA)
Brief Title: The Influence of Raltegravir on Pravastatin Pharmacokinetics(GRAPPA)
Acronym: GRAPPA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Dr. D.M. Burger, hospital pharmacist, Radboud University Nijmegen Medical Centre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UMCN-AKF 07.05
Record Dates: First submitted 2008-04-23; First posted 2008-04-24 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2011-05

CONDITIONS: HIV Infections
Keywords: interaction; statins; pharmacokinetics
MeSH Terms: conditions — HIV Infections | interventions — Pravastatin; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): Pravastatin 40 mg QD for 4 days
  Interventions: Drug: Pravastatin
- B (Active Comparator): Raltegravir 400mg BD for 4 days
  Interventions: Drug: Raltegravir
- C (Experimental): Interaction between pravastatin and raltegravir
  Interventions: Drug: Pravastatin and raltegravir

INTERVENTIONS:
Drug: Pravastatin — 40 mg tablet; QD; 4 days
  Other Names: Selektine
  Arms: A
Drug: Raltegravir — 400mg tablet; BD 4 days
  Other Names: Isentress
  Arms: B
Drug: Pravastatin and raltegravir — pravastatin 40mg tablet QD for 4 days; raltegravir 400mg tablet BD for 4 days
  Other Names: Selektine and Isentress
  Arms: C

SUMMARY:
The purpose of this trial is to determine the effect of raltegravir on pravastatin pharmacokinetics and vice versa by intrasubject comparison.

DETAILED DESCRIPTION:
Pravastatin is a first choice statin for HIV-infected patients. Therefore, raltegravir and pravastatin are expected to be co-administered frequently in HIV-infected patients.Since both agents share the same metabolic pathway, there is a potential for a pharmacokinetic drug-drug interaction.

Because co-administration will be indicated in many HIV-infected patients, it is essential to investigate this potential interaction.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 and not older than 55 years of age.
* Subject does not smoke more than 10 cigarettes, 2 cigars, or 2 pipes per day.
* Subject has a Quetelet Index (Body Mass Index) of 18 to 30 kg/m2.
* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
* Subject is in good age-appropriate health condition.
* Subject has a normal blood pressure and pulse rate.

Exclusion Criteria:

* Documented history of sensitivity/idiosyncrasy to medicinal products or exci-pients.
* Positive HIV test.
* Positive hepatitis B or C test.
* Pregnant female or breast-feeding female.
* Therapy with any drug.
* Relevant history or presence of pulmonary disorders (especially COPD), car-diovascular disorders, neurological disorders (especially seizures and mi-graine), gastro-intestinal disorders, renal and hepatic disorders, hormonal disorders (especially diabetes mellitus), coagulation disorders.
* Fasting triglyceride levels > 8.0 mmol/L
* Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
* History of or current abuse of drugs, alcohol or solvents.
* Inability to understand the nature and extent of the trial and the procedures required.
* Participation in a drug trial within 60 days prior to the first dose.
* Donation of blood within 60 days prior to the first dose.
* Febrile illness within 3 days before the first dose

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-05; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of pravastatin and raltegravir. | t=0 (predose), 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 10, 12 and (24: for pravastatin only) hours post ingestion on Days 4, 18 and 32. Trough level on Day 2, 16 and 30.

SECONDARY OUTCOMES:
To investigate the non-steady state changes in serum low density lipoprotein (LDL) cholesterol secondary to pravastatin use in the presence or absence of raltegravir | Screening and Days 1, 5, 15, 19, 29 and 33.
Determination of pharmacokinetic parameters | at each sampling time
To evaluate the safety of combined use of pravastatin and raltegravir | entire trial

CONTACTS AND LOCATIONS:
Overall Officials: David M Burger, PharmD PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Result] van Luin M, Colbers A, van Ewijk-Beneken Kolmer EW, Verweij-van Wissen CP, Schouwenberg B, Hoitsma A, da Silva HG, Burger DM. Drug-drug interactions between raltegravir and pravastatin in healthy volunteers. J Acquir Immune Defic Syndr. 2010 Sep;55(1):82-6. doi: 10.1097/QAI.0b013e3181d9a354. PMID 20395869
- See also: Publication in Journal of Acquired Immune Deficiency Syndromes; Issue: Volume 55(1), 1 September 2010, pp 82-86 — http://www.ncbi.nlm.nih.gov/pubmed/20395869